CLINICAL TRIAL: NCT02139241
Title: The Efficacy and Safety of Ramosetron in Patients Undergoing Off Pump Coronary Artery Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Ramosetron_opcab
Record Dates: First submitted 2013-11-12; First posted 2014-05-15 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2014-05

CONDITIONS: Coronary Artery Bypass Graft Triple Vessel; Hypotension
MeSH Terms: conditions — Hypotension | interventions — ramosetron; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ramosetron (Experimental): Intravenous administration of ramosetron 0.3 mg before the induction of general anesthesia
  Interventions: Drug: Ramosetron
- Control (Placebo Comparator): Intravenous administration of 2ml normal saline before the induction of general anesthesia
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ramosetron — 0.3 mg IV as bolus before induction of general anesthesia
  Other Names: Nasea
  Arms: Ramosetron
Drug: Normal saline — 2 ml normal saline as bolus before induction of general anesthesia
  Arms: Control

SUMMARY:
The purpose of this study is to assess the effects of ramosetron on corrected QT interval in patients undergoing off pump coronary artery bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective off-pump coronary artery bypass graft surgery

Exclusion Criteria:

* Emergency operation
* preoperative use of any inotropics or mechanical assist device
* severe liver disease (>Child class II)
* dialysis dependent renal failure
* Left ventricular ejection fraction <30 %
* Combined major surgery like carotid endarterectomy
* Previous allergy history to any 5-hydroxytryptamine type 3 (5-HT3) antagonist
* Preoperative QT prolongation ( 500 >msec) or arrhythmia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2013-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
corrected QT interval (QTc interval) | up to 240 minutes after induction of general anesthesia
  at 1,2,3,5,10,15,30,45,60,90,120,240 minutes after ramosetron injection, at the time of operation end, ICU 12hour

SECONDARY OUTCOMES:
hypotension or bradycardia during the peri-induction period and the coronary anastomosis period | up to 240 minutes after induction of general anesthesia
incidence of postoperative atrial fibrillation | during the hospital stay (from ICU admission to hospital discharge, average of 1 week)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Havrilla PL, Kane-Gill SL, Verrico MM, Seybert AL, Reis SE. Coronary vasospasm and atrial fibrillation associated with ondansetron therapy. Ann Pharmacother. 2009 Mar;43(3):532-6. doi: 10.1345/aph.1L544. Epub 2009 Mar 3. PMID 19261954
- [Background] Sahoo T, SenDasgupta C, Goswami A, Hazra A. Reduction in spinal-induced hypotension with ondansetron in parturients undergoing caesarean section: a double-blind randomised, placebo-controlled study. Int J Obstet Anesth. 2012 Jan;21(1):24-8. doi: 10.1016/j.ijoa.2011.08.002. Epub 2011 Nov 18. PMID 22100822
- [Derived] Kim TK, Cho YJ, Lim CW, Min JJ, Choi EK, Hong DM, Jeon Y. Effect of ramosetron on QTc interval: a randomised controlled trial in patients undergoing off-pump coronary artery bypass surgery. BMC Anesthesiol. 2016 Aug 3;16(1):56. doi: 10.1186/s12871-016-0222-1. PMID 27488394